CLINICAL TRIAL: NCT04004650
Title: Gluteal Turnover Flap for Closure of the Perineal Wound After Abdominoperineal Resection for Rectal Cancer
Acronym: BIOPEX2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Gijsbert Musters, MD PhD, reseach coordinator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL65461.018.18
Record Dates: First submitted 2019-06-10; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Wound Heal; Abdominoperineal Resection; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary closure (No Intervention): Primary perineal closure after extralevator abdomino perineal resection
- Gluteal turnover flap (Experimental): Gluteal flap reconstruction of the pelvic floor after extralevator abdomino perineal resection
  Interventions: Procedure: Gluteal turnover flap

INTERVENTIONS:
Procedure: Gluteal turnover flap — Link to procedure: https://www.youtube.com/watch?v=u7_vH2_1ZZc
  Arms: Gluteal turnover flap

SUMMARY:
Background:

About 700 patients per year undergo an abdominoperineal resection (APR) for distal rectal cancer (Dutch Colorectal Audit 2016).Neoadjuvant (chemo)radiotherapy is often used to further improve locoregional control. Morbidity after APR is substantial and mainly consisting of perineal wound problems in about 35% of the patients. lf primary healing of the perineal wound after APR doesn't occur, secondary healing can take up to one year, and there is even a small proportion of patients in whom a chronic perineal wound or fistula persists after one year. During this long period, intensive wound care is necessary. This results in a heavy burden on both patient and health care resources.

Objective:

The high morbidity rate of the perineal wound has resulted in a continuing discussion on how to close the perineal defect after APR. Our research group recently published the BIOPEX-study (NL42094.018.12), in which 104 patients were randomized between primary perinea! wound closure and biological mesh closure of the pelvic floor after APR with preoperative radiotherapy for rectal cancer. Similar uncomplicated perineal wound healing rate at 30 days (Southampton wound score < 2) was found: 63% versus 66%, respectively. The hypothesis behind this negative trial result is related to the perineal dead space between the skin and the biological mesh. Fluid will accumulate in this dead space with the risk of secondary contamination and abscess formation, leading to wound dehiscence and purulent discharge. Autologous tissue flaps have been suggested to improve perineal wound healing based on several cohort studies. At least in the Netherlands, these flaps are used only for selected patients with the large defects and highest risk of wound problems, because of the more extensive surgery with added surgical trauma and operative time, and associated donor site morbidity. For these reasons, primary perineal closure (control arm of BIOPEX) is still the standard of care in the Netherlands.

A gluteal turnover flap (GT flap) is a small transposition flap trom the unilateral adjacent perineal skin and subcutaneous fat, which is flipped into the perineal dead space, and stitched with the de-epithelialised dermis to the contralateral pelvic floor remnant. Subsequently, the perineal subcutaneous fat and skin are closed over the flap in the midline, thereby not adding a donor site scar. A small pilot study trom our group showed that this is a promising solution for routine perineal closure after APR.

Study design:

In this multicenter single blinded study, eligible patients will be randomized between pelvic floor reconstruction using a GT flap (intervention arm) and primary closure of the perineal defect (standard arm). The perineal wound healing will be evaluated at 14 days and 1, 3, and 6 months post-operatively using the Southampton wound scoring system by an independent observer.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of primary rectal cancer or recurrent rectal cancer
* scheduled for abdominalperineal resection
* older then 18 years

Exclusion Criteria:

* intersphincteric APR
* (biological) mesh placement
* extended resections (sacral resection except for coccyx resection, (posterior) exenteration)
* severe systemic diseases affecting wound healing except diabetes (i.e. renal failure requiring dialysis, liver cirrhosis, and immune compromised status like HIV), collagen disorders (i.e. Marfan)
* enrolment in other trials with overlapping primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Perineal wound healing rate 30 days | 30 days
  The primary endpoint of the study is the percentage of uncomplicated perineal wound healing defined as a Southampton wound score of less than Il at 30 days postoperatively.

SECONDARY OUTCOMES:
Perineal wound healing | 14 days, 3 and 6 months postoperatively
  Southampton wound score
Re-intervention or re-admission rate | 1,3,6 months
  Need tor re-intervention or re-admission related to pre-sacral abscess or either perineal wound problems.
Perineal hernia rate | 1,3,6 months
  lncidence of symptomatic and asymptomatic perineal hernia
Health-related quality of life | 1,3,6 months
  questionnaires: The 5-level EQ-5D version (EQ-5D-5L)
Quality of Life in cancer patients | 1,3,6 months
  questionnaires: European Organization for Research and Treatment for Cancer Quality of Life Questionnaire (C30-QL2, CR29)
Generic quality of Life | 3,6 months
  questionnaires: Short Form Survey (SF36)
Urogenital Distress | 1,3,6 months
  questionnaires: Urogenital Distress Inventory (UDI-6)
Incontinence scale | 1,3,6 months
  questionnaires:Incontinence Impact Questionnaire short form (IIQ-7)
Urogenital function | 1,3,6 months
  questionnaires: international index of erectile function (IIEF)
Female sexual distress | 1,3,6 months
  questionnaires: Female sexual distress scale (FSDS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Tanis, Prof. MD. Phd, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreisel SI, Sharabiany S, Tuynman J, Belgers EHJ, Singh B, Chaudhri S, van Geloven AAW, Vuylsteke RJCLM, de Wilt JHW, Melenhorst J, Leijtens JWA, Vermaas M, Rothbarth J, Verhoef C, Burger JWA, Polat F, Fabry HFJ, Aalbers AGJ, Wijsman JH, Lamme B, van der Bilt JDW, Lapid O, van Dieren S, Hompes R, Tanis PJ, Musters GD. Perineal Wound Closure Using Gluteal Turnover Flap After Abdominoperineal Resection for Rectal Cancer: The BIOPEX-2 Randomized Clinical Trial. JAMA Surg. 2025 Apr 1;160(4):378-385. doi: 10.1001/jamasurg.2024.6818. Erratum In: JAMA Surg. 2025 Apr 1;160(4):471. doi: 10.1001/jamasurg.2025.0523. PMID 39908025
- [Derived] Sharabiany S, Blok RD, Lapid O, Hompes R, Bemelman WA, Alberts VP, Lamme B, Wijsman JH, Tuynman JB, Aalbers AGJ, Beets GL, Fabry HFJ, Cherepanin IM, Polat F, Burger JWA, Rutten HJT, Bosker RJI, Talsma K, Rothbarth J, Verhoef C, van de Ven AWH, van der Bilt JDW, de Graaf EJR, Doornebosch PG, Leijtens JWA, Heemskerk J, Singh B, Chaudhri S, Gerhards MF, Karsten TM, de Wilt JHW, Bremers AJA, Vuylsteke RJCLM, Heuff G, van Geloven AAW, Tanis PJ, Musters GD. Perineal wound closure using gluteal turnover flap or primary closure after abdominoperineal resection for rectal cancer: study protocol of a randomised controlled multicentre trial (BIOPEX-2 study). BMC Surg. 2020 Jul 23;20(1):164. doi: 10.1186/s12893-020-00823-7. PMID 32703182